CLINICAL TRIAL: NCT06409767
Title: Impact of an Early Warning System on the Prognosis of Patients With Hematological Malignancies Receiving Intensive Chemotherapy With or Without Hematopoietic Cell Transplantation, a Multicenter Cluster Randomized Study
Brief Title: Impact of an Early Warning System on the Prognosis of Patients With Hematological Malignancies Receiving Intensive Chemotherapy With or Without Hematopoietic Cell Transplantation.
Acronym: ALHERT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 49RC23_0425; ID-RCB (Other: ANSM)
Record Dates: First submitted 2024-05-07; First posted 2024-05-10 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Leukemia; Lymphoma; Multiple Myeloma
Keywords: Intensive chemotherapy; hematopoietic cell transplantation; early ICU admission
MeSH Terms: conditions — Leukemia; Lymphoma; Multiple Myeloma

STUDY DESIGN:
Intervention Model Description: Cluster randomized trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interventional arm (Experimental)
  Interventions: Other: Real-time calculation of the NEWS with ICU admission if NEWS ≥ 7.
- Control arm (No Intervention)

INTERVENTIONS:
Other: Real-time calculation of the NEWS with ICU admission if NEWS ≥ 7. — The calculation of NEWS requires vital signs such as respiratory rate, peripheral oxygen saturation, need for oxygen therapy, body temperature, arterial pressure, heart rate, and level of consciousness. Each parameter used to calculate the NEWS will be collected least three times a day by the attending nurse.
  Arms: Interventional arm

SUMMARY:
Patients with hematologic malignancies requiring intensive chemotherapy are at risk for life-threatening complications. Organ failure may appear rapidly and delay in initiating life-sustaining interventions may result in increased mortality. This encourages great alertness although not all patients require close monitoring. It is therefore critical to identify which patients are the most at risk for clinical deterioration to consider increased surveillance in these patients. The benefit of early intensive care unit (ICU) admission, as soon as the first signs of organ dysfunction appear, must also be clarified. Such an intervention could increase survival of patients by close monitoring and early initiation of organ-specific interventions but could also be responsible for anxiety and increased use of ICU resources.

Many teams have analyzed the impact of early warning systems (EWS) including vital signs to detect organ dysfunction early on. It has been shown that these EWS could positively impact survival in many medical fields (pre-hospital, medicine or surgery departments). A few retrospective studies have explored the impact of EWS in hematology, with overall good prediction for ICU admission and mortality. Until now, it has however not been formally demonstrated that early ICU admission, as soon as the first signs of organ dysfunction appear, could benefit patients with hematologic malignancies. A randomized controlled trial studying the impact of early intervention would clarify the role of such a strategy.

In this study, the investigators will prospectively evaluate the implementation of the National Early Warning Score (NEWS), with systematic referral to the ICU in high-score patients, to improve the survival of patients receiving intensive chemotherapy in ten academic centers. This score is one of the most performant and most frequently used to predict organ failure. Its calculation only requires vital signs such as respiratory rate, peripheral oxygen saturation, need for oxygen therapy, body temperature, arterial pressure, heart rate, and level of consciousness. The investigators will therefore study the impact of ICU admission in patients with high NEWS in a randomized, controlled trial. A cluster randomization is planned in which the centers will be randomized between usual care (control group) and interventional care with transfer to the ICU in the event of a NEWS score ≥7 (interventional group). Each parameter used to calculate the NEWS will be collected at least three times a day by the attending nurse.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient
* Hospitalization in a protected unit of a hematology department for induction therapy of acute myeloid leukemia or acute lymphoblastic leukemia induction, intensive chemotherapy with autologous hematopoietic cell transplantation, allogeneic hematopoietic cell transplantation
* Expected length of stay in the hematology department of at least 7 days
* Patient with social security
* Signed informed consent form

Exclusion Criteria:

* Decision of care limitation with decision not to transfer to ICU or not initiate organ support
* Pregnant, parturient or breastfeeding woman
* Person deprived of liberty by judicial or administrative decision
* Person under forced psychiatric care
* Person under legal protection
* Person unable to express consent
* Hospitalization for Chimeric Antigenic Receptor (CAR) T-cell therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2224 (Estimated)
Dates: Start 2025-04-10 (Actual); Primary Completion 2028-04-11 (Estimated); Study Completion 2028-07-11 (Estimated)

PRIMARY OUTCOMES:
In-hospitality mortality and/or inition of organ support | 3 months
  In-hospital mortality and/or initiation of organ support (invasive mechanical ventilation, vasopressors [Epinephrin, Dobutamine or Adrenaline], renal replacement therapy, extracorporeal circulation [ECMO]).

SECONDARY OUTCOMES:
Relative weight of each parameter used to calculate the NEWS for predicting the risk of organ failure requiring life-sustaining organ support | 3 months
  Cox proportional hazards model with shared fragility to explain the occurrence over time of one or more organ support. The model's explanatory variables will be the different parameters used to calculate the NEWS.
Feasibility of implementing early warning scores in routine practice | 3 months
  Proportion of patients with NEWS ≥7 effectively admitted to the ICU in the investigational arm.
To assess quality of life of patients according to treatment arm. | 3 months
  Quality of life scores measured by the EQ-5D-5L questionnaire at days 0, 30, and 90 will be analyzed using linear mixed models (LMM) to account for repeated measures, for both the overall score and each dimension (mobility, self-care, usual activities, pain/discomfort, and anxiety/depression).
economic evaluation | 3 months
  Cost-utility analysis will estimate the incremental cost utility ratio (ICUR) in cost per quality-adjusted life year (QALY) gained and cost-effectiveness analysis will estimate the incremental cost effectiveness ratio (ICER) in cost per life year gained.

CONTACTS AND LOCATIONS:
Locations (10):
- France (10):
  - Centre Hospitalier Amiens-Picardie, Amiens
  - Centre Hospitalier Universitaire d'Angers, Angers
  - Centre Hospitalier Universitaire Besancon, Besançon
  - Centre Hospitalier Universitaire Brest, Brest
  - Centre Hospitalier universitaire Nancy, Nancy
  - Centre Hospitalier Universitaire Nantes, Nantes
  - Centre Hospitalier Universitaire poitiers, Poitiers
  - centre Hospitalier Universitaire Saint etienne, Saint-Etienne
  - centre Hospitalier Universitaire Strasbourg, Strasbourg
  - centre Hospitalier Universitaire Tours, Tours

IPD SHARING:
Plan to Share IPD: No